CLINICAL TRIAL: NCT05844202
Title: A Phase 1 Open-label, Active-controlled, Randomized Dose-finding Study to Evaluate Safety, Tolerability, and Immunogenicity of Intradermal and Subcutaneous Application of the Plasmid DNA SARS-CoV-2 Omicron BA.2 Vaccine Alveavax-v1.2 in Primary Ad26.COV2.S Vaccinated Healthy Individuals
Brief Title: Safety, Tolerability and Immunogenicity of Alveavax-v1.2, a BA.2/Omicron-optimized, DNA Vaccine for COVID-19 Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvea Holdings, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Alvea-VAX-P00001; DOH-27-062022-5157 (Registry Identifier: SANCTR)
Record Dates: First submitted 2023-05-02; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Sars-CoV-2 Infection
Keywords: Sars; Sars-CoV-2; COVID-19; Vaccine; pDNA; plasmid DNA; COVID19
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low dose (Experimental): 0.5 mg Alveavax-v1.2 in one ID injection
  Interventions: Drug: Alveavax-v1.2
- Standard dose (Experimental): 2 mg Alveavax-v1.2 in one ID injection
  Interventions: Drug: Alveavax-v1.2
- High dose (Experimental): 8mg Alveavax-v1.2 in four ID injections
  Interventions: Drug: Alveavax-v1.2
- Comparator (Active Comparator): 0.5ml Janssen Ad26.COV2.S COVID-19 vaccine in one IM injection
  Interventions: Drug: Janssen Ad26.COV2.S
- Subcutaneous (Experimental): 8mg Alveavax-v1.2 in one SC injection
  Interventions: Drug: Alveavax-v1.2

INTERVENTIONS:
Drug: Alveavax-v1.2 — BA.2/Omicron optimized plasmid DNA vaccine for the prevention of COVID-19
  Other Names: Alveavax
  Arms: High dose; Low dose; Standard dose; Subcutaneous
Drug: Janssen Ad26.COV2.S — COVID-19 vaccine by Janssen / Johnson & Johnson
  Other Names: Janssen
  Arms: Comparator

SUMMARY:
The investigated product is a Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Booster Vaccine candidate optimized for the Omicron/BA.2 variant. There are currently no licensed, variant-optimized vaccines to prevent infection with SARS-CoV-2 Omicron/BA.2. Approved or authorized SARS-CoV-2 vaccines are expensive, require a stringent cold chain, and have large-scale manufacturing issues, resulting in very limited availability in low- and middle-income countries (LMICs). Given the rapid global spread of the Omicron/BA.2 variant and potential for future novel SARS-CoV-2 variants, the rapid development of an easy-to-manufacture and easy-to-distribute vaccine is of great importance.

The objective of the study is to assess the tolerability, safety, and immunogenicity of different doses and routes of administration of the Alveavax-v1.2 vaccine in healthy individuals.

The study aims to evaluate:

* the safety and tolerability of Alveavax-v1.2 in healthy participants compared to a control booster vaccine in a dose-finding design;
* the immunogenicity against SARS-CoV-2 BA.2/Omicron after a booster dose of Alveavax-v1.2;
* the clinical efficacy against SARS-CoV-2 after a booster dose of Alveavax-v1.2;
* and the success rate of intradermal (ID) injections.

DETAILED DESCRIPTION:
This is a first in human, open-label, active-controlled, randomized dose-finding study to evaluate safety, tolerability, and immunogenicity of intradermal (ID) and subcutaneous (SC) application of the plasmid DNA SARS-CoV-2 Omicron BA.2 vaccine Alveavax-v1.2 in primary Ad26.COV2.S vaccinated healthy individuals.

Primary Ad26.COV2.S vaccinated participants will be randomized into one of 5 treatment arms to receive Alveavax-v1.2 or a Ad26.COV2.S control booster vaccine.

Participants will be enrolled at multiple sites in South Africa within 28 days after the initial screening to ensure they meet all the inclusion criteria and none of the exclusion criteria.

Each participant will be administered a booster vaccine on Day 1 of the study and will be monitored afterwards. Solicited local/systemic reactions will be recorded after vaccination in the participant's diary card for up to 7 days (the vaccine administration day and 6 days later).

A total of 130 participants of any sex, aged between 18 and 65 years, who satisfy the inclusion and exclusion criteria are planned to be enrolled in five groups and with vaccine administered according to their dose arm as follows:

Low dose: 0.5 mg Alveavax-v1.2 in one ID injection

Standard dose: 2 mg Alveavax-v1.2 in one ID injection

High dose: 8mg Alveavax-v1.2 in four ID injections

SC injection: 8mg Alveavax-v1.2 in one SC injection

Control: Janssen Ad26.COV2.S in one intramuscular (IM) injection

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and female volunteers between 18 and 65 years of age, inclusive.
2. Participants who received a primary Janssen Ad26.CoV2.S vaccine ≥ 60 days prior to receiving the study vaccine.
3. Body mass index within the range 18 - 32 kg/m2 both inclusive.
4. Participants who, judged by the Investigator, are in stable health as determined by their pre-study medical history, physical examination, and clinical laboratory tests.
5. Female participants must be either of non-childbearing potential, i.e., surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year postmenopausal; or, if of childbearing potential, they must be abstinent or have used adequate contraceptive precautions for 30 days prior to receiving the study vaccination and 84 days post-vaccine.
6. Sexually active male participants who are considered sexually fertile must agree to use a barrier method of contraception during sexual activity with a female of childbearing potential from the time of vaccination until at least 84 days after the vaccination.
7. Participants must provide written informed consent or their legal representative must understand and give written consent to the procedure.
8. Participants must be willing and able to comply with all the required study visits and follow-up required by this protocol, and be able to complete the diary card after vaccination or have a caregiver available to assist with these matters.

Exclusion Criteria:

1. Received any other SARS-CoV-2 vaccination than a single Janssen Ad26.COV2.S vaccine or plans to receive any additional SARS-CoV-2 vaccination within 90 days after the study vaccine (Day 1).
2. Recovered from SARS-CoV-2 infection determined by history of a positive SARS-CoV-2 test (e.g. PCR, rapid antigen test, etc.) or suspicion of a SARS-CoV-2 infection based on the (verbal) medical history within less than 60 days from the day of vaccination (Day 1) in this study.
3. History of close contact (face-to-face contact within 1 meter or contact in a closed space for more than 15 minutes) without wearing a face-mask with a confirmed active SARS-CoV-2-positive patient within 5 days prior to Day 1.
4. Have received any live-virus vaccine within 4 weeks or inactivated vaccine, including influenza vaccine, within 2 weeks (both licensed and investigational vaccines) prior to the study vaccine (Day 1).
5. Previous participation in any clinical trial of a SARS-CoV-2 vaccine candidate.
6. Have any febrile illness (temperature ≥ 38°C/100.4°F) or any active acute illness or infection (including a positive SARS-CoV-2 PCR test) within 7 days prior to administration of vaccination (Day 1) in this study. Participants may be re-evaluated once all symptoms have resolved.
7. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) or contraindications to any component of the study intervention(s).
8. History of, or positive screening test for human immunodeficiency virus I or II.
9. Any clinically significant finding during screening or check-in that, in the Investigator's judgment, results in an increased safety risk.
10. History of cerebral venous sinus thrombosis, antiphospholipid syndrome, or a history of heparin-induced thrombocytopenia and thrombosis (HITT or HIT type 2).
11. Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 3 months, except topical and inhaled steroids, or short-term oral steroids (course lasting ≤14 days or ≤20 mg/day).
12. History of receiving blood transfusion, blood products, immunoglobulin, or immune stimulants within 3 months prior to Day 1.
13. Is currently participating in any other study or has received any investigational drug in the last 6 weeks or 5× the half-life of the drug (whichever is longer) prior to screening.
14. For female participants of childbearing potential who are pregnant (positive pregnancy test at the screening or check-in), currently breastfeeding, or attempting to conceive.
15. Any addiction that may interfere with the participant's ability to comply with trial procedures.
16. Inability to be venipunctured or tolerate venous, IM, SC, or ID puncture.
17. Have a rash, dermatological condition, tattoo, or any other abnormality at the injection site that may interfere with injection site reaction rating. Investigator discretion will be permitted with this exclusion criterion.
18. Use of prophylactic medications (e.g., antihistamines [H1 receptor antagonists], nonsteroidal anti-inflammatory drugs [NSAIDs], systemic glucocorticoids, non-opioid and opioid analgesics) within 24 hours prior to the vaccination to prevent or pre-empt symptoms due to vaccination.
19. Any condition or abnormal baseline findings or any other unspecified reason, which in the Investigator's judgment might increase the risk to the participant or decrease the chance of obtaining satisfactory data needed to achieve the objective of the study.
20. Participants identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator, or employee with direct involvement in the proposed study, or any employees of the Sponsor company.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Alveavax-v1.2 in healthy participants compared to a control booster vaccine (Day 7) | Day 7
  The overall number of participants and incidence proportion of any solicited local and systemic AEs within seven days of dose administration
Safety and tolerability of Alveavax-v1.2 in healthy participants compared to a control booster vaccine (Day 28) | Day 28
  The overall number of participants and incidence proportion of unsolicited adverse events (AEs) within 28 days of dose administration
Safety and tolerability of Alveavax-v1.2 in healthy participants compared to a control booster vaccine | Day 168
  The overall number of participants and incidence of serious adverse events (SAEs), adverse events of special interest (AESIs), and AEs leading to participant discontinuation throughout the trial

SECONDARY OUTCOMES:
Immunogenicity as humoral immune response against SARS-CoV-2 BA.2/Omicron after a booster dose of Alveavax-v1.2 | Day 28
  Geometric Mean Titer (GMT) and change in GMT of SARS-CoV-2 BA.2 binding antibodies
Success rate of intradermal injections | Day 1
  Absolute number and fraction of ID injections which generated a ≥ 1 mm and ≥ 7 mm in diameter clearly demarcated bleb, clearly visible for at least 20 seconds, for 0.5 mg and 2 mg Alveavax-v1.2 respectively

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — TASK
Locations (8):
- South Africa (8):
  - JOSHA Research, Bloemfontein, Free State
  - NMMM Pharmmedica Health and Clinical Research, Johannesburg, Gauteng
  - MERC Kempton Park, Kempton Park, Gauteng
  - Ubuntu Clinical Research Center, Krugersdorp, Gauteng
  - Ubuntu Clinical Research Center Lenasia, Lenasia, Gauteng
  - Setshaba Research Centre, Soshanguve, Gauteng
  - MERC Research Pty Ltd, Middelburg, Mpumalanga
  - TASK applied Science Brooklyn Chest Hospital, Ysterplaat, Western Cape